CLINICAL TRIAL: NCT06816706
Title: Comparison of Physiological Effects of Two Types of High-Flow Tracheal Oxygen Versus T-Piece During Spontaneous Breathing Trials in Mechanically Ventilated Patients
Brief Title: Comparison of Physiological Effects of Two High-Flow Tracheal Oxygen Versus T-Piece During Spontaneous Breathing Trials
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jian-Xin Zhou (Other)
Responsible Party: Sponsor-Investigator, Jian-Xin Zhou, Professor, Capital Medical University
Organization: Capital Medical University (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IIT2024-157-002
Record Dates: First submitted 2025-02-04; First posted 2025-02-10 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-02

CONDITIONS: Critical Care; Oxygen Therapy; Mechanical Ventilation
Keywords: high-flow tracheal oxygen; T piece; spontaneous breathing trial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Modified high flow tracheal oxygen-40L/min (Experimental): Modified high-flow tracheal oxygen with a flow rate of 40L/min will be performed in mechanically ventilated patients undergoing spontaneous breathing trials.
  Interventions: Procedure: Modified high flow tracheal oxygen-40L/min
- Standard high flow tracheal oxygen-40L/min (Experimental): Standard high-flow tracheal oxygen with a flow rate of 40L/min will be performed in mechanically ventilated patients undergoing spontaneous breathing trials.
  Interventions: Procedure: Standard high flow tracheal oxygen-40L/min
- T-piece (Experimental): T-piece will be performed in mechanically ventilated patients undergoing spontaneous breathing trials.
  Interventions: Procedure: T-piece
- Modified high-flow tracheal oxygen-60L/min (Experimental): Modified high-flow tracheal oxygen with a flow rate of 60L/min will be performed in mechanically ventilated patients undergoing spontaneous breathing trials.
  Interventions: Procedure: Modified high-flow tracheal oxygen-60L/min
- Standard high-flow tracheal oxygen-60L/min (Experimental): Standard high-flow tracheal oxygen with a flow rate of 60L/min will be performed in mechanically ventilated patients undergoing spontaneous breathing trials.
  Interventions: Procedure: Standard high-flow tracheal oxygen-60 L/min

INTERVENTIONS:
Procedure: Modified high flow tracheal oxygen-40L/min — Modified high-flow tracheal oxygen with a flow rate of 40L/min will be performed.
  Arms: Modified high flow tracheal oxygen-40L/min
Procedure: Standard high flow tracheal oxygen-40L/min — Standard high-flow tracheal oxygen with a flow rate of 40 L/min will be performed.
  Arms: Standard high flow tracheal oxygen-40L/min
Procedure: T-piece — T-piece will be performed.
  Arms: T-piece
Procedure: Modified high-flow tracheal oxygen-60L/min — Modified high-flow tracheal oxygen with a flow rate of 60L/min will be performed.
  Arms: Modified high-flow tracheal oxygen-60L/min
Procedure: Standard high-flow tracheal oxygen-60 L/min — Standard high-flow tracheal oxygen with a flow rate of 60 L/min will be performed.
  Arms: Standard high-flow tracheal oxygen-60L/min

SUMMARY:
Spontaneous breathing trials (SBT) are essential for assessing extubation tolerance, yet optimal approaches are debated. High-flow nasal oxygen offers benefits like precise oxygen delivery, flow-related positive end-expiratory pressure generation and improved lung function. While high-flow tracheal oxygen can also be used as an SBT method, it has reduced physiological effects due to bypassing the upper airway with a more open circuit. To enhance this limitation, investigators developed a modified high-flow tracheal oxygen tube with a smaller expiratory end diameter to increase expiratory resistance and airway pressure. This is a prospective randomized crossover study that aims to compare the physiological effects of standard and modified high-flow tracheal oxygen versus T-piece during SBT.

DETAILED DESCRIPTION:
A spontaneous breathing trial (SBT) is a crucial step in the weaning and extubation process for assessing extubation tolerance. However, the optimal approach for conducting SBTs remains a topic of debate.

High-flow nasal oxygen has been shown to provide several physiological benefits, including precise control of the fraction of inspired oxygen, generation of flow-related positive end-expiratory pressure, increased end-expiratory lung volume, improved oxygenation, and enhanced carbon dioxide elimination. High-flow oxygen therapy can also be applied via an artificial airway as high-flow tracheal oxygen. Previous studies have identified this therapy as a potential alternative for SBTs. However, compared to high-flow nasal oxygen, high-flow tracheal oxygen exhibits significantly diminished physiological effects due to the bypassing of the narrow nasopharynx, glottis, and upper airway as well as a more open circuit.

To address this limitation, the investigators have developed a modified high-flow tracheal oxygen tube with a reduced expiratory end tube diameter. This modification aims to create higher expiratory resistance and airway pressure, thereby simulating the physiological effects of HFNC. This study is a prospective randomized crossover physiological study designed to compare the effects of standard and modified high-flow tracheal oxygen versus T-piece during spontaneous breathing trials. Key physiological parameters will be assessed, including airway pressure, end-expiratory lung volume, vital signs, oxygenation, and respiratory workload.

ELIGIBILITY:
Inclusion Criteria:

1. Mechanical ventilation for more than 24 hours
2. Considered by the physicians for the readiness to wean and ready for spontaneous breathing trials

Exclusion Criteria:

1. Age younger than 18 years old
2. Pregnancy
3. Hemodynamic instability (mean arterial pressure <60 mmHg, heart rate >140 or <60 bpm)
4. Respiratory and oxygenation instability (respiratory rate > 35bpm or oxygen saturation measured by pulse oximetry <90%)
5. Neuromuscular diseases or phrenic nerve injury
6. Recent trauma or surgery to the trachea, esophagus, neck, chest, or stomach
7. Pneumothorax or placement of a chest drainage
8. Contraindication to electrical impedance tomography (EIT) (implantable defibrillator)
9. Anticipating withdrawal of life support

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Mean expiratory airway pressure | From enrollment to the end of treatment at 4 hours
  Mean expiratory airway pressure will be measured during standard and modified high-flow tracheal oxygen versus T-piece.
Positive end-expiratory pressure | From enrollment to the end of treatment at 4 hours
  Positive end-expiratory pressure will be measured during standard and modified high-flow tracheal oxygen versus T-piece.
Change of end-expiatory lung volume | From enrollment to the end of treatment at 4 hours
  Change of end-expiatory lung volume will be measured during standard and modified high-flow tracheal oxygen versus T-piece.

SECONDARY OUTCOMES:
Respiratory rate | From enrollment to the end of treatment at 4 hours
  Respiratory rate will be measured during standard and modified high-flow tracheal oxygen versus T-piece.
Tidal volume | From enrollment to the end of treatment at 4 hours
  Tidal volume will be measured during standard and modified high-flow tracheal oxygen versus T-piece.
End-tidal carbon dioxide | From enrollment to the end of treatment at 4 hours
  End-tidal carbon dioxide will be measured during standard and modified high-flow tracheal oxygen versus T-piece.
Pulse oxygen saturation | From enrollment to the end of treatment at 4 hours
  Pulse oxygen saturation will be measured during standard and modified high-flow tracheal oxygen versus T-piece.
Esophageal pressure-time product | From enrollment to the end of treatment at 4 hours
  Esophageal pressure-time product will be measured during standard and modified high-flow tracheal oxygen versus T-piece.
Tidal swing of esophageal pressure | From enrollment to the end of treatment at 4 hours
  Tidal swing of esophageal pressure will be measured during standard and modified high-flow tracheal oxygen versus T-piece.
Respiratory muscle pressure | From enrollment to the end of treatment at 4 hours
  Respiratory muscle pressure will be measured during standard and modified high-flow tracheal oxygen versus T-piece.
Dynamic transpulmonary pressure | From enrollment to the end of treatment at 4 hours
  Dynamic transpulmonary pressure will be measured during standard and modified high-flow tracheal oxygen versus T-piece.

CONTACTS AND LOCATIONS:
Overall Officials: Jian-Xin Zhou, MD, PhD, Principal Investigator — Capital Medical University
Locations (1):
- Beijing Shijitan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xu SS, Zhang RZ, An X, Miao MY, Wang YF, Li HL, Zhou JX. Physiological effects of high-flow oxygen via endotracheal tube versus T-piece strategies during spontaneous breathing trials: a study protocol and statistical analysis for a single-centre randomised crossover study. BMJ Open. 2025 Sep 16;15(9):e105360. doi: 10.1136/bmjopen-2025-105360. PMID 40962338